CLINICAL TRIAL: NCT00159263
Title: Effect of Symbicort on GR (Glucocorticoid Receptor) Translocation in Induced Sputum in Comparison With Budesonide, Formoterol and Placebo. A Single Dose Exploratory Study in Patients With Mild Asthma
Brief Title: Effect of Symbicort on GR Localisation in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BU-039-0005
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Asthma
Keywords: Asthma; Glucocorticoid; Long-acting beta2-adrenoceptor; Inhaled corticosteroids
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebos
- Formoterol (Experimental): Oxis(®) 12 μg
  Interventions: Drug: Formoterol Inhalant Powder
- Budesonide low dose (Experimental): Pulmicort(®) 200 μg
  Interventions: Drug: Budesonide Powder
- Budesonide high dose (Experimental): Pulmicort(®) 800 μg
  Interventions: Drug: Budesonide Powder
- Budesonide/formoterol combination single (Experimental): single 100/6 μg SYM100
  Interventions: Drug: Budesonide and Formoterol Product
- Budesonide/formoterol combination double (Experimental): double 200/12 μg SYM200
  Interventions: Drug: Budesonide and Formoterol Product

INTERVENTIONS:
Drug: Placebos — Dry powder inhaler
  Arms: Placebo
Drug: Formoterol Inhalant Powder — 12ug
  Other Names: Oxis
  Arms: Formoterol
Drug: Budesonide Powder — Inhaler
  Other Names: Pulmicort
  Arms: Budesonide high dose; Budesonide low dose
Drug: Budesonide and Formoterol Product — Combination Inhaler, Symbicort
  Other Names: Combination Inhaler, Symbicort
  Arms: Budesonide/formoterol combination double; Budesonide/formoterol combination single

SUMMARY:
To investigate a possible interaction between formoterol and budesonide on GR-translocation and to compare the effect of different doses of Symbicort (80/4.5 and 2x80/4.5 mcg) with the effect of budesonide (200 mcg and 800 mcg) on GR translocation, and to investigate the effect of the study drugs on exhaled NO (bronchial and alveolar fraction.

DETAILED DESCRIPTION:
Combination therapy with inhaled corticosteroids (ICS) and long-acting β(2)-adrenergic agonists (LABA) is reported to have superior effects on controlling asthma symptoms to ICS alone; however, there is no molecular-based evidence to explain the clinical effects. Here, the effect of the ICS/LABA combination was compared with ICS on glucocorticoid receptor (GR) activation in sputum macrophage.

In a randomised, double-blind cross-over placebo-controlled 6-visit study, 10 patients with mild asthma were given placebo, formoterol (Oxis(®) 12 μg), budesonide (Pulmicort(®) 200 μg :BUD200, or 800 μg :BUD800), or budesonide/formoterol combination (Symbicort(®)) as a single 100/6 μg (SYM100) or double 200/12 μg (SYM200) dose. Sputum macrophages were separated by plate adhesion from induced sputum. GR binding to the glucocorticoid-response elements on oligonucleotides (GR-GRE binding) was evaluated by ELISA. mRNA expression of MAP-kinase phosphatase (MKP)-1 and IL-8 were measured by quantitative RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild steroid-naïve asthma (ATS criteria) of either sex with FEV1 >70 % pred
* Able to produce sputum after sputum induction
* Exhaled NO (flow 50 ml/s) ≥ 20 ppb
* Written informed consent

Exclusion Criteria:

* Current upper respiratory tract infections
* Use of inhaled and/or oral GCS within 4 weeks prior to visit 1
* Treatment with antileukotrienes, theophylline, tiotropium and ipratropium within 2 weeks prior to screening visit
* Hypersensitivity to any of the investigational drugs or lactose
* Use of any beta blocking agent (including eye-drops)
* Women who are pregnant, breast-feeding or planning a pregnancy during the study. Women must be postmenopausal (at least one year must have passed after the last menstruation), surgically sterile or using acceptable contraceptives, as judged by the investigator
* Any significant disease or disorder (e.g. cardiovascular, pulmonary (other than asthma), gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subjects ability to participate in the study
* Inability to tolerate temporary withdrawal of bronchodilatory therapy
* Subjects not considered capable, as judged by the investigator, of following instructions of the study, e.g. because of a history of alcohol or drug abuse or any other reason
* Previous randomization in this study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Essilfie-Quaye S, Ito K, Ito M, Kharitonov SA, Barnes PJ. Comparison of Symbicort(R) versus Pulmicort(R) on steroid pharmacodynamic markers in asthma patients. Respir Med. 2011 Dec;105(12):1784-9. doi: 10.1016/j.rmed.2011.08.020. Epub 2011 Sep 7. PMID 21903370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10patient recruited mild asthma
Groups:
- Placebo: first intervention is placebo, then Formoterol, then Budesonide low dose, then Budesonide high dose, then Budesonide/Formoterol single, then Budesonide/Formoterol double
- Formoterol: First intervention is formoterol, then placebo, then Budesonide low dose, then Budesonide high dose, then Budesonide/Formoterol single, then Budesonide/Formoterol double
- Budesonide Low Dose: First intervention is Budesonide low dose, then placebo, then Formoterol, then Budesonide high dose, then Budesonide/Formoterol single, then Budesonide/Formoterol double
- Budesonide High Dose: First intervention is Budesonide high dose, then placebo, then Formoterol, then Budesonide low dose, then Budesonide/Formoterol single, then Budesonide/Formoterol double
- Budesonide/Formoterol Single: First intervention is Budesonide/Formoterol single, then placebo, then Formoterol, then Budesonide low dose, then Budesonide high dose, then Budesonide/Formoterol double
- Budesonide/Formoterol Double: First intervention is Budesonide/Formoterol double, then placebo, then Formoterol, then Budesonide low dose, then Budesonide high dose, then Budesonide/Formoterol single
Period: First Intervention
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Intervention
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Sixth Intervention
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Crossover study, same volunteers in all arm, received the following interventions: formoterol, Budesonide low and high dose, or combination of these
Arm/Group | Overall Study
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in GR-GRE Binding
Description: The GR-GRE binding is the glucocorticoid receptor (GR) DNA binding affinity. GR-GRE activity as assed by enzyme-immunosorbent assay
Time Frame: 1-2h
Population: Crossover, each patient had all treatments
Measure: Median (Inter-Quartile Range); unit: GRE activity (OD)
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Combination Single | Budesonide/Formoterol Combination Double
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
GRE activity (OD) | 1.4 [0.5 to 2] | 1.4 [0.3 to 2.6] | 1.6 [0.7 to 2.0] | 2.3 [1.1 to 7] | 3.5 [1.3 to 6.1] | 3 [1.5 to 6]
Statistical Analysis 1: Comparison: Placebo vs Budesonide/Formoterol Combination Single; Test type: Other — Friedman ANOVA followed Dunn's pairwise comparisons; p = 0.04, ANOVA

2. Primary Outcome: Changes in MKP-1 mRNA
Description: Changes in MKP-1 mRNA measured by PCR
Time Frame: 1-2h
Measure: Median (Inter-Quartile Range); unit: MKP1/GNB2L1 ratio
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Combination Single | Budesonide/Formoterol Combination Double
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
MKP1/GNB2L1 ratio | 1 [0.1 to 1] | 3 [1 to 44] | 3 [2 to 70] | 4 [4 to 51] | 5 [3 to 150] | 5 [3 to 150]
Statistical Analysis 1: Comparison: Placebo vs Budesonide/Formoterol Combination Double; Test type: Other — Friedman Anova; p = 0.01, ANOVA

3. Primary Outcome: IL8 mRNA
Description: Measured by PCR
Time Frame: 1-2h
Measure: Median (Inter-Quartile Range); unit: IL8/GNB2L1 ratio
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Combination Single | Budesonide/Formoterol Combination Double
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
IL8/GNB2L1 ratio | 1 [0.1 to 1.7] | 4 [0.1 to 20] | 4 [0.1 to 20] | 0.4 [0.1 to 1.3] | 0.2 [0.1 to 0.7] | 0.2 [0.1 to 1.4]
Statistical Analysis 1: Comparison: Placebo vs Budesonide/Formoterol Combination Double; Test type: Other — Friedman Anova; p = 0.04, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo: Patients who received placebo treatment
- Formoterol: Patients who received Formoterol treatment
- Budesonide Low Dose: Patients who received Budesonide low dose treatment
- Budesonide High Dose: Patients who received Budesonide high dose treatment
- Budesonide/Formoterol Single: Patients who received Budesonide/Formoterol single dose treatment
- Budesonide/Formoterol Double: Patients who received Budesonide/Formoterol double dose treatment
Arm/Group | Placebo | Formoterol | Budesonide Low Dose | Budesonide High Dose | Budesonide/Formoterol Single | Budesonide/Formoterol Double
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes